CLINICAL TRIAL: NCT04345562
Title: Cesarean Section Skin Prep - Does Skin Preparation Pattern Affect Skin Bacterial Burden
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Megan Piacquadio, Principal Investigator, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2019-165
Record Dates: First submitted 2020-03-09; First posted 2020-04-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cesarean Section Complications; Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back and forth pattern (Active Comparator): Abdominal skin prep using ChloraPrep 2 x 26 mL single use applicators. The first applicator will be applied to the skin prep over the suspected skin incision site for 30 sec - the first applicator will then be used in a back and forth pattern work up towards the upper edge of the surgical field. The first applicator will then be discarded. The second applicator will then again start at the expected site of the incision and again working inferiority until the lower edge of the surgical field is reached.
  Interventions: Procedure: Skin preparation patterns with ChloraPrep 2 x 26 mL single
- Circular pattern (Active Comparator): Abdominal skin prep using ChloraPrep 2 x 26 mL single use applicators. The first applicator will be applied to the skin over the suspected skin incision site for 30 sec - the applicator will then be moved in a circular pattern moving outwards form the incision site until approximately half of thee surgical field is cleaned. The second applicator will then be used to complete the surgical prep until the entire surgical field is prepped in accordance with the package instructions.
  Interventions: Procedure: Skin preparation patterns with ChloraPrep 2 x 26 mL single

INTERVENTIONS:
Procedure: Skin preparation patterns with ChloraPrep 2 x 26 mL single — 2 different patterns of skin preparation
  Other Names: ChloraPrep 2 x 26 mL single use applicators

SUMMARY:
Currently there is no study investigating best skin cleaning patterns prior to cesarean deliveries. As a result, doctors perform skin preparation using random unstudied techniques. Techniques vary from Hospital to Hospital and even within the same institution. The most widely used topical skin preparation is ChloraPrep and the manufacturer has not recommended a specific pattern to be used in order to abdominally prep prior to C-sections. In addition most studies do not examine the effectiveness in the obese population. The manufacture has established a recommended dosage area of 13in x13in per ChloraPrep stick as well as timing from initial preparation until the practice reached its maximum antiseptic benefit.

Our current cesarean infection rate is very low, at just 1.6% over the last 12 months (September 2107-2018). This is significantly lower than the average cesarean section infection rate in the United States which is around 7.4% using iodine based preparations. Cesarean deliveries are one of the most common major surgeries performed in the United States, 31.9% of all births are by cesarean section. The risk of infection following a cesarean delivery is nearly 5 times that of a vaginal delivery. However, there is still no study that examines the pattern which ChloraPrep is applied to the abdomen prior to a cesarean delivery in patients with a BMI greater than 30. The pattern of skin preparation appears to be heavily related to physician training and personal bias.

DETAILED DESCRIPTION:
Currently there is no study investigating optimal skin preparations patterns prior to cesarean deliveries. As a result, there are many practitioners that perform skin preparation, cleaning of the surgical site, using random unstudied patterns. Patterns vary from Hospital to Hospital and even within the same institution. The most widely used topical skin preparation is ChloraPrep and the manufacturer has not recommended a specific pattern to be used in order to abdominally prep prior to C-sections. They have published data instructing one on the surface area for which a ChloraPrep stick is verified to be used for as well as timing from initial preparation until the cleaner has reached its maximum antiseptic benefit.

Our current cesarean infection rate is 1.6% over the last 12 months (September 2107-2018). This is significantly lower than the average cesarean section infection rate in the United States which is estimated to be around 7.4%.[i] Cesarean deliveries are one of the most common major surgeries performed in the united states, 31.9% of all births are by cesarean section.[ii] The risk of infection following a cesarean delivery is nearly 5 times that of a vaginal delivery[iii]. However, there is still no study that examines the pattern which ChloraPrep, the most widely used skin cleaner, is applied to the abdomen prior to a cesarean delivery.

There is currently no study that looks at pattern of skin preparation prior to cesarean section. The manufacture simply recommends gentle scrubbing. The pattern of skin preparation appears to be related to your training.

This study aims to look at topical skin preparation patterns prior to cesarean section. As a proxy for likelihood of infection the investigators will collect data on surface bacterial burden prior to incision but after abdominal prep is complete as well as post surgically. The assumption is that if there is a significant skin burden postoperatively that one method of skin preparation is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital for scheduled C-section.
2. C-section incision must be Pfannenstiel
3. Preoperative antibiotics administered in accordance with ACOG recommendations
4. BMI >30

Exclusion Criteria:

1. Patient is currently on immunosuppression therapy.
2. Patient is allergic to any medications or materials used during the research study
3. BMI >45 are excluded
4. Patient refuses to participate in the study.
5. Case is converted from plan to stat cesarean section
6. Age less than 18
7. If patient is determined to be unable to be consented

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Skin bacterial burden | 1-4 days
  Culture bacterial burden prior to incision

SECONDARY OUTCOMES:
Surgical site infection | 4 weeks
  Culture diagnosis of surgical site infections
Hospital Re-admissions | 4 weeks
  All cause hospital readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piacquadio, DO, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share data with other researchers